CLINICAL TRIAL: NCT06687291
Title: Cognitive Impact Associated With Surgery For Gastric Or Esophageal Cancer
Acronym: CASE
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Lampi, Principal Investigator, Karolinska Institutet
Other Study IDs: Ethical approval 2024-00971-01
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Gastroesophageal Cancer (GC); Postoperative Delirium (POD); Quality of Life (QOL); Frailty; Malnutrition; Sarcopenia; Chemobrain; Chemotherapy; Depression
Keywords: postoperative delirium; gastroesophageal cancer; Frailty; Quality of life; Preoperative depression; Malnutrition; Sarcopenia; Chemobrain; Chemotherapy
MeSH Terms: conditions — Emergence Delirium; Frailty; Malnutrition; Sarcopenia; Chemotherapy-Related Cognitive Impairment; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants identified with postoperative delirium: Participants identified with postoperative delirium will be asked (at the routine follow-up meeting after surgery) to participate in an qualitative interview in order to understand the participant's experience of postoperative delirium.
- CASE-study participants: All included participants in the CASE-study.
  * The assessment of cognitive function will be performed using the validated 4AT Test (4AT). Cognitive impact will be assessed at baseline before neoadjuvant chemotherapy (if chemotherapy is indicated) and at patient admission for surgery, postoperative day 1, 3 and 7, and at follow-up 4-8 weeks after surgery.
  * Risk factors for POD will be explored by investigate the relationship between postoperative delirium, chemotherapy preoperative depression, frailty, quality of life, malnutrition and sarcopenia. Patients will report health-related quality of life using the validated EORTC QLQC-C30 and EORTC QLQ-OG25 questionnaires. Frailty and depression will be measured preoperatively with Clinical Frailty Scale (CFS-9) and the Patient Health Questionnaire (PHQ-9). Malnutrition is evaluated by using Patient-Generated Subjective Global Assessment (PG-SGA). Sarcopenia is assessed through CT-scan, which is conducted as part of clinical routine.

SUMMARY:
The primary objective of this observational study is to investigate the incidence of Post Operative Delirium (POD) after gastroesophageal cancer surgery. Secondary objectives are to investigate the relationship between POD, preoperative depression, frailty, quality of life, malnutrition and sarcopenia.

Participants identified with POD will be asked (at the routine follow-up meeting after surgery) to participate in an qualitative interview, in order to understand the participant's experience of postoperative delirium.

The main objective aims to answer:

What is the incidence of POD after gastroesophageal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with esophageal or gastric cancer, treated with (or without) chemotherapy and surgery.
* Age ≥18 at the time for inclusion.
* Participate on a voluntary basis and can (for any reason) end its participation during the study.
* Capable of giving informed consent.

Exclusion Criteria:

* Patients with preoperative cognitive dysfunction such as dementia.
* Patients who are inoperable due to metastases.
* Patients unable to communicate due to severely impaired hearing and/or - seeing.
* Patients with ongoing drug and/or alcohol abuse.
* Patients who cannot give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with esophageal or gastric cancer who will be treated with (or without) chemotherapy and surgery at Karolinska University Hospital in Huddinge (Sweden).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2027-11-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | From enrollment to the follow up meeting after surgery, approximate 6 months.
  The assessment of cognitive function will be performed using the validated 4AT Test (4AT).
  Cognitive impact will be assessed at baseline before neoadjuvant chemotherapy (if chemotherapy is indicated) and at patient admission for surgery, postoperative day 1, 3 and 7, and at follow-up 4-8 weeks after surgery.

SECONDARY OUTCOMES:
Preoperative depression | From enrollment to admission for surgery
  A risk factor for postoperative delirium is preoperative depression. Depression will be measured preoperatively with the Patient Health Questionnaire (PHQ-9).
Preoperative frailty | At admission for surgery
  Frailty is a risk factor for post operative delirium. Frailty will be measured preoperatively with Clinical Frailty Scale (CFS-9).
Health-related quality of life | From enrollment to the follow up meeting after surgery, approximate 6 months.
  Low score in quality of life is a risk factor for delirium. Patients will report health-related quality of life using the validated European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQC-C30) and EORTC validated Quality of Life Questionnaire for Oesophago-Gastric cancer (QLQ-OG25).
Malnutrition | At admission for surgery
  Patients with malnutrition before surgery have a higher risk of developing post-operative delirium. Malnutrition is assessed by using Patient-Generated Subjective Global Assessment (PG-SGA) before surgery.
Sarcopenia | From enrollment to admission for surgery
  There is association between preoperative sarcopenia and postoperative delirium in patients undergoing gastrointestinal cancer surgery. Sarcopenia is assessed by using CT-scan in clinical routine.

OTHER OUTCOMES:
Patients experience of Postoperative delirium | The interview takes place 2 weeks after follow up-meeting
  All participants that suffered from POD will be invited to participate in an interview, with a maximum number of 25 participants. A semi-structured one-on-one interview with the aim to describe patient experiences of POD will be used. The semi-structured interview technique allows the interviewer to ask probing questions for clarification when necessary. An interview guide will be used to ensure covering issues such as cognition, memory loss, attention, awareness and orientation to the environment. The participant will be asked for participation at the follow-up meeting after surgery. The interview takes place 2 weeks after follow up-meeting after surgery at the location (or via that media) that best serve the participant. The interview will be recorded and transcribed, then analysed using qualitative content analysis with an inductive and latent approach.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lampi, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tieges Z, Maclullich AMJ, Anand A, Brookes C, Cassarino M, O'connor M, Ryan D, Saller T, Arora RC, Chang Y, Agarwal K, Taffet G, Quinn T, Shenkin SD, Galvin R. Diagnostic accuracy of the 4AT for delirium detection in older adults: systematic review and meta-analysis. Age Ageing. 2021 May 5;50(3):733-743. doi: 10.1093/ageing/afaa224. PMID 33951145
- [Background] Liu J, Li J, Wang J, Zhang M, Han S, Du Y. Associated factors for postoperative delirium following major abdominal surgery: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2023 Jun;38(6):e5942. doi: 10.1002/gps.5942. PMID 37260053
- [Background] Loh KP, Janelsins MC, Mohile SG, Holmes HM, Hsu T, Inouye SK, Karuturi MS, Kimmick GG, Lichtman SM, Magnuson A, Whitehead MI, Wong ML, Ahles TA. Chemotherapy-related cognitive impairment in older patients with cancer. J Geriatr Oncol. 2016 Jul;7(4):270-80. doi: 10.1016/j.jgo.2016.04.008. Epub 2016 Jul 5. PMID 27197918
- [Background] Hughes CG, Boncyk CS, Culley DJ, Fleisher LA, Leung JM, McDonagh DL, Gan TJ, McEvoy MD, Miller TE; Perioperative Quality Initiative (POQI) 6 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Postoperative Delirium Prevention. Anesth Analg. 2020 Jun;130(6):1572-1590. doi: 10.1213/ANE.0000000000004641. PMID 32022748
- See also: Cognitive test 4AT — https://www.the4at.com/
- See also: European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQC-C30). Quality of life questionnaire for patients with cancer. — https://ki.se/media/253910/download
- See also: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Oesophago-Gastric cancer (QLQ-OG25) questionnaire. Quality of life questionnaire for patients with gastroesophageal cancer. — https://www.eortc.org/app/uploads/sites/2/2018/08/Specimen-OG25-English.pdf
- See also: Patient Health Questionnaire (PHQ-9), questionnaire about depression — https://viss.nu/download/18.668ca5111744c9a9eed82aaf/1610623941602/PHQ-9_svensk.pdf
- See also: Clinical Frailty Scale (CFS-9). Frailty questionnaire — https://janusinfo.se/download/18.54c15e0616f53615ae5882fd/1578400633984/Clinical-Frailty-Scale-svensk.pdf
- See also: Patient-Generated Subjective Global Assessment (PG-SGA). A validated tool for screening and assessing malnutrition — https://pt-global.org/wp-content/uploads/2024/02/PG-SGA-Metric-version-4.3.20-std-logo-SWE.pdf